CLINICAL TRIAL: NCT03086213
Title: the Safety and Effectiveness of the Effects on the Perioperative Pain Control Comparing Between the Thoracic Paravertebral Nerve Block Using the Camera Guided and the Intrathoracic Intercostals Nerve Block for the Management of Nonintubated Local Regional Analgesia in Uniport Thoracoscopic Surgery for the Undetermined Solitary Nodules Patients
Brief Title: Comparative Study of Nonintubated Uniport Thoracoscopic Surgery Using Thoracic Paravertebral Nerve Block Versus Intercostal Nerve Block for Peripheral Solitary Pulmonary Nodule Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Third People's Hospital (Other)
Responsible Party: Principal Investigator, xia zhaohua, Director, Head of thoracic surgical department, Principal investigator, Associate clinical professor, Shenzhen Third People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19800911
Record Dates: First submitted 2017-03-07; First posted 2017-03-22 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Solitary Pulmonary Nodule or Tuberculoma
Keywords: nonintubated uniport thoracoscopic surgery; paravertebral nerve block; intercostal nerve block; peripheral solitary pulmonary nodule
MeSH Terms: conditions — Tuberculoma | interventions — Propofol; Sufentanil; Dexmedetomidine; Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paravertebral nerve block group (Experimental): non-intubated thoracic paravertebral nerve block of regional anesthesia Thoracic paravertebral nerve block of regional anesthesia at the T4 thoracic interspace
  Interventions: Drug: Propofol; Drug: Sulfentanyl; Drug: Dexmedetomidine; Drug: Lidocaine; Drug: Ropivacaine
- intercostals nerve block group (Active Comparator): non-intubated intercostal nerve block of regional anesthesia Thoracic intercostal nerve block of regional anesthesia at the T3/4/5 thoracic interspace
  Interventions: Drug: Propofol; Drug: Sulfentanyl; Drug: Dexmedetomidine; Drug: Lidocaine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Propofol — anaesthetic
Drug: Sulfentanyl — anaesthetic
Drug: Dexmedetomidine — anaesthetic
Drug: Lidocaine — local anaesthetics
Drug: Ropivacaine — local anaesthetics

SUMMARY:
The aim of this study is to study the safety and effectiveness of the effects on the perioperative pain control comparing between the thoracic paravertebral nerve block using the camera guided and the intrathoracic intercostals nerve block for the management of nonintubated local regional analgesia in uniport thoracoscopic surgery for the undetermined solitary nodules patients.

DETAILED DESCRIPTION:
Thoracoscopic minor lung resection has been the reasonable option for the diagnosis and treatment of management of the undetermined peripheral pulmonary nodules. Uniport procedure could reduce postoperative pain score, the length of hospital stay, moreover, nonintubated technique can avoid the disadvantages of conventional general anesthesia such as ventilator induced lung injury, sore throat or voice change. The nonintubated technique without tracheal intubation under spontaneous ventilation combined with uniport or single port thoracoscopic surgery has emerged as the least invasive procedure of wedge resection of peripheral pulmonary nodules, even the anatomical thoracoscopic lobectomy along with mediastinal lymph nodule dissection in case of the diagnosis of the primary lung cancer during the operation.

The initial experience of nonintubated thoracoscopic surgery included the intravenous controlled sedation and pain , thoracic epidural analgesia and thoracic vagus nerve block, due to series of adverse events of the epidural analgesia, operator was willing to perform the intrathoracic intercostal nerve block guided by camera during the operation and was considered as the simple and safety method for regional analgesia .However, the intercostal nerve block can not employ the adequate pain control ,after the surgery, the patient controlled analgesia is as usual needed.

The previous study showed that paravertebral block was the same effect on relieved pain as thoracic epidural analgesia and had the less complications such as hypotension, nausea or vomiting. With the advance in the technique of application of ultrasound, it is more interesting that using the ultrasound technique before the surgery is performed for the adequate pain control of the local regional analgesia in nonintubated surgery under spontaneous ventilation. However, ultrasound technique is difficult to have the skilled experience for the most anaesthetists and increase the related puncture complications such as hematoma, bleeding or pneumothorax. The method used study is guided by camera which is very simple and safety by avoidance of the puncture of the partial pleura or intercostal blood vessel, The investigators once used this approach for postoperative pain control under general intubation for lung cancer patients, so the investigators have had a skilled experience for achieving regional analgesia of nonintubated uniport thoracoscopic wedge resection.

So far, there has been no articles about thoracic paravertebral nerve block for regional analgesia of nonintubated thoracoscopic procedure patients. The investigators designed the study to compare the short term outcome on thoracic paravertebral nerve block in nonintubated technique with those of intercostal nerve block in uniport nonintubated video-assisted thoracoscopic surgery(VATS) as the control group.

This study will be performed at the third people's hospital of Shenzhen. A total of 48 patients will be enrolled(24 patients in each arms).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* the undetermined peripheral solitary pulmonary nodule or tuberculoma was enrolled
* the well cardiopulmonary function
* age between 18 and 65 years old
* less airway secretion
* body mass index less than 25
* I to II grade of the American Society of Anesthesiologists
* no metabolic diseases

Exclusion Criteria:

* refusal or inability to comply with the informed consent
* the nodule of the nature of the non small cell lung caner is excluded
* hypovolemia, blood disorders or abnormal clotting mechanism
* the abnormal cardiopulmonary function(the American Society of Anesthesiologists greater than 3)
* lower airway infection,more than airway secretion
* abnormal anatomy of the spine,the history of thoracic back surgery
* impaired lung function(forced expiratory volume in second 1 less than predicted), or asthma uncontrolled on medications
* constrained cardiac output such as hypertrophic cardiomyopathy, mitral stenosis or complete atrioventricular block
* extensive pleural adhesion
* overweight (body mass index no less than 25)
* difficulty airway
* chronic pain score more than 5 before the surgery
* the history of bilateral thoracotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- the Third People's Hospital of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data available to other researcher.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Per Arm: paravertebral nerve block and intercostal nerve block
Arm/Group | Per Arm
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: there is two arms for the overall subjects divided into the two different regional anesthesia.
  years
    PVB: number analyzed (Participants) | 24
    PVB | 34.6 (10.47)
    INB: number analyzed (Participants) | 24
    INB | 42.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: there is two arms for the overall subjects of this study divided into the two different regional anesthsia
  Participants
    PVB: Female | 30
    PVB: Male | 18
    INB: Female | 30
    INB: Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Comparing the Inflammatory Markers During the Operation After the Intervention of the Each Group
Description: serum concentrations of Interleukin-6
Time Frame: During the operation, an average of one hour
Measure: Mean (Standard Deviation); unit: pg/L
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Number analyzed (Participants) | 24 | 24
pg/L
  Interleukin-6 T0 | 33 (8) | 35 (8)
  Interleukin-6 T1 | 39 (10) | 42 (9)
  Interleukin-6 T2 | 44 (9) | 53 (11)
  Interleukin-6 T3 | 47 (9) | 54 (13)
Statistical Analysis 1: Comparison: Paravertebral Nerve Block Group vs Intercostals Nerve Block Group; null hypothesis; Test type: Non-Inferiority — the definition of non-inferiority analysis is that the new method is no less effective than standard interventions; p = 0.025, t-test, 2 sided — whether or not the p-value is adjusted for multiple comparisons and the a priori threshold for statistical significance; degrees of freedom; Mean Difference (Final Values) = 10, 95% CI 2-sided [5 to 95], Standard Deviation 0.025 — Paravertebral nerve block arm represents the numerator and intercostal block represents the denominator for relative risk

2. Primary Outcome: Concentration of Cortisol at Different Point During the Operation
Time Frame: During the operation, an average of one hour
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Number analyzed (Participants) | 24 | 24
ng/mL
  During the operation, 0m | 120 (31) | 125 (33)
  During the operation, 15m | 208 (49) | 221 (66)
  During the operation, 30m | 258 (69) | 290 (71)
  During the operation, 60m | 267 (77) | 318 (74)
Statistical Analysis 1: Comparison: Intercostals Nerve Block Group; null hypothesis; Test type: Superiority — During the calculation of sample size,a sample size of 24 patients per group was calculated as being required to ensure 90% power of detecting the difference-if any-as statistically significant at the 5% level; p < 0.05, t-test, 2 sided — the p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance; degrees of freedom is defined as sample size subtraction one

3. Secondary Outcome: Comparing the Hemodynamics of the Intervention of the Each Group During the Operation
Description: data of mean arterial pressure
Time Frame: During the operation, an average of one hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Number analyzed (Participants) | 24 | 24
mmHg
  mean arterial pressure T0 | 79 (7) | 80 (8)
  mean arterial pressure T1 | 85 (8) | 86 (8)
  mean arterial pressure T2 | 72 (9) | 85 (7)
  mean arterial pressure T3 | 78 (6) | 80 (8)

4. Secondary Outcome: Comparing the Hemodynamics of the Intervention of the Each Group During the Operation
Description: data of heart rate
Time Frame: During the operation, an average of one hour
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Number analyzed (Participants) | 24 | 24
bpm
  heart rate T0 | 78 (7) | 79 (7)
  heart rate T1 | 84 (6) | 85 (7)
  heart rate T2 | 81 (8) | 92 (9)
  heart rate T3 | 78 (7) | 80 (5)

5. Secondary Outcome: Comparing the Blood Gas Analysis After the Intervention of the Each Group
Description: data of arterial partial pressure of oxygen(PaO2) and PaCO2 at different point during the operation
Time Frame: During the operation, an average of one hour
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Number analyzed (Participants) | 24 | 24
cmH2O
  arterial partial pressure of oxygen(PaO2) | 95.2 (1.8) | 96.2 (1.8)
  arterial partial pressure of PaC | 51.1 (11.1) | 47.3 (9.7)
Statistical Analysis 1: Comparison: Intercostals Nerve Block Group; null hypothesis; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.05, t-test, 2 sided; Degree of freedom is defined as sample size subtraction one

6. Secondary Outcome: Number of Participants With Puncture Related Complications
Description: puncture related complications
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
Number analyzed (Participants) | 20 | 20
Participants
  hematoma | 2 | 3
  pain of punture position | 2 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Paravertebral Nerve Block Group | Intercostals Nerve Block Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paravertebral Nerve Block Group (N=24) | Intercostals Nerve Block Group (N=24)
bleeding related to the puncture in the pleural cavity (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03086213/SAP_000.pdf
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03086213/Prot_001.pdf
  • Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03086213/ICF_002.pdf